CLINICAL TRIAL: NCT04229927
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of BPDO-1603 in Patients With Moderate-to-severe Alzheimer's Disease
Brief Title: BPDO-1603 Intervention Trial in Patients With Moderate-to-severe Alzheimer's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-007-04
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-01

CONDITIONS: Moderate-to-severe Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BPDO-1603
- Arm 2 (Placebo Comparator)
  Interventions: Drug: BPDO-1603

INTERVENTIONS:
Drug: BPDO-1603 — Arm1 : 1 tablet of the test drug, and 1 tablet of placebo reference drug
  Arm2 : 1 tablet of the reference drug, and 1 tablet of placebo test drug

SUMMARY:
A multicenter, randomized, double-blind, active-controlled, phase III clinical trial to evaluate the efficacy and safety of BPDO-1603 in patients with moderate-to-severe Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* A voluntary, written informed consent from the patient or the patient´s representative.
* Male or female patients ≥ 45 years of age as of the date of informed consent.
* Diagnosed with probable AD according to the National Institute on Aging-Alzheimer's Association [NIA-AA (2011)] criteria.
* MMSE score of ≥ 5 and ≤ 20 during screening period.
* CDR-GS of 2 ~ 3 or GDS of 4 ~ 7 during screening period.
* Ongoing cholinesterase inhibitor therapy with stable dose of 10 mg/day donepezil hydrochloride for more than 12 weeks (inclusive) prior to screening, and can continue this therapy until randomization without any change in the dosage regimen of donepezil hydrochloride.

Exclusion Criteria:

* Magnetic resonance imaging (MRI) or computed tomography (CT) findings obtained within the past 12 months (ie, 48 weeks) from screening or at screening, as a cause of dementia other than probable AD.
* History of other organic disease, such as vascular dementia, CNS infections (e.g., human immunodeficiency virus [HIV], syphilis), head injury, Creutzfeldt-Jakob disease, Niemann-Pick's disease, Huntington's disease, Parkinson's disease, epilepsy, or stroke.
* Evidence of other neurological disorders which include seizure disorder that may interfere with the patient's cognition or ability to perform the study procedures.
* Use of Memantine Hydrochloride within 1 month prior to screening

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in SIB total scores | from baseline to Week 24
CIBIC-plus total score | at Week 24 (Baseline score will be from CIBIS

CONTACTS AND LOCATIONS:
Overall Officials: Seonghye CHOI, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea